CLINICAL TRIAL: NCT04795557
Title: Effect of ADAPT232 Supplementation on Recovery of Patients in Rehabilitation Period in Long COVID-19: a Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Efficacy of Adaptogens in Patients With Long COVID-19
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Swedish Herbal Institute AB (Industry)
Collaborators: National Family Medicine Training Centre, Georgia (Unknown); Tbilisi State Medical University (Other); Phytomed AB (Other)
Responsible Party: Principal Investigator, Alexander Panossian, Head of Research and Development at Phytomed AB, Phytomed AB
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHIRD-2021-01; Nr2-2021/86 (Registry Identifier: Biomedical Research Ethics Committee)
Record Dates: First submitted 2021-03-08; First posted 2021-03-12 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Covid19
Keywords: Long Covid; fatigue; headache; attention disorder,; depression; anxiety
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome; Fatigue; Headache; Cognition Disorders; Depression; Anxiety Disorders | interventions — ADAPT 232

STUDY DESIGN:
Intervention Model Description: Patients will be randomized in a manner of 1:1 for study drug (ADAPT-232) and Standard of Care to Placebo and Standard of Care.
  Patient treatment period will last 2 weeks. During this time, patients will be monitored for adverse events.
  There will be a follow up period in order to check adverse events and study drug efficacy
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ADAPT232 (Experimental): 50 patients take ADAPT-232® oral solution in the daily dose of 60 ml ( 30 ml two times daily) for 14 days.
  One mL of oral solution contains:
  Schisandra chin. fructus native extract 10,0 mg DERnative 2,0-5,0:1 Eleutherococcus sent. radix native extract 2,6 mg DERnative 17-30:1 Rhodiola rosea radix native extract. 3,0 mg DERnative 2,0-5,0:1 Inactive excipients,
  Interventions: Dietary Supplement: ADAPT-232 oral solution
- Placebo (Placebo Comparator): 50 patients take Placebo oral solution in the daily dose of 60 ml ( 30 ml two times daily) for 14 days.
  Interventions: Other: Placebo oral solution

INTERVENTIONS:
Dietary Supplement: ADAPT-232 oral solution — One ml of ADAPT 232/CHISAN oral solution contains:
  Fructus Schizandrae native extract DERnative 2-4:1, (extraction solvent . 95% ethanol) - 10 mg corresponding to 20-40 mg dried fruit; Radix Eleutherococci native extract DERnative 17-30:1 (extraction solvent - 70% ethanol) - 2.6 mg corresponding to 44-78 mg dried rhizomes, and Radix Rhodiolae native extract DERnative 2-5:1 (extraction solvent - 70% ethanol) - 3 mg corresponding to 6-30 mg dried rhizomes.
  Excipients
  Other Names: Chisan
  Arms: ADAPT232
Other: Placebo oral solution — Excipients
  Arms: Placebo

SUMMARY:
The aim of this clinical trial of a fixed combination of standardized extracts from Rhodiola rosea roots, Schisandra chinensis berry and Eleutherococcus senticosus root (ADAPT-232) in COVID-19 patients is to demonstrate possible efficacy of adjuvant treatment with ADAPT-232 in decreasing the duration of the convalescence, alleviation of fatigue, headache, attention deficit, difficult and rapid respiration, depression, anxiety and other symptoms of Long COVID-19 during rehabilitation period.

DETAILED DESCRIPTION:
Rationale. Currently, numerous clinical trials on efficacy antiviral preparations in COVID-19 patients are in progress, however little is known on effective treatment of comorbid complications or COVID long-haulers during convalescence, particularly on fatigue, headache, attention deficit, and depression. The aim of this study is to assess eficacy of an adaptogenic preparation ADAPT-232 on recovery of COVID-19 Patients in rehabilitation period after discharge from Intensive Care Units.

Pathogenesis and progression of COVID-19 is multistep process, which requires correct therapeutic strategy on various steps of initiation of overall defense response to pathogen and its resolution. Consequently, effective prevention or treatment of COVID-19 requires pharmaceutical corrections of many components innate, adaptive immune system, phases I-III metabolizing enzymes of detoxifying and repair systems as well as on the SARS-Cov-2 virus' life cycle and proliferation. We suggest that It can be achieved by multitarget pharmaceutical intervention of herbal preparations that have polyvalent and pleiotropic actions on host defence systems, like adaptogens, which are known as natural stress-protective compounds or plant extracts that increase adaptability, resilience, and survival of organisms. In this context, complex mixtures of natural compounds (or herbal extracts) synergistically targeting multiple elements of molecular networks involved in inflammatory defence response are presumably more effective than the monodrugs, targeting only one receptor.

Adaptogenic preparations were tested in controlled clinical trials for the treatment of common cold and associated uncomplicated upper respiratory infections as well as for the prevention of common colds. The studies confirm their safety and efficacy presumably due to antiviral, anti-inflammatory and adaptogenic activity. Further studies are required to evaluate their efficacy in COVID-19 and other viral respiratory invidious diseases.

One more possible benefit of adaptogens in COVID-19 might be their beneficial effect during convalescence of patents. This indication for use is based on the results of a randomized, placebo controlled double blind study of Chisan/ADAPT-232 (a fixed combination of three adaptogenic plants Eleutherococcus senticosus - Rhodiola rosea and Schisandra chinensis) in pneumonia. The results obtained in that study clearly indicate that adjuvant treatment of pneumonia patients with Chisan (ADAPT-232) significantly decreases the period of antibiotic therapy required for recovery, decreasing the duration of the acute phase of the illness, and improves the mental performance of patients during the convalescence period with an accompanying improvement in the quality-of-life.

ADAPT 232® is a formulation used in different dosage forms for the enhancement of mental and physical capacities in case of tiredness or during convalescence. Chisan (ADAPT-232) has been on the Swedish market as a natural remedy since 1979.

Approved indications:

Sweden: Herbal medicinal product used as an adaptogen in case of decreased performance such as fatigue and sensation of weakness.

Denmark: Herbal medicinal product for fatigue and re-convalescence Canada: Herbal medicine for the enhancement of mental and physical capacities in case of tiredness or during convalescence

Recruitment:

Individuals will be recruited by doctors of National Family Medicine Training Centre (NFMTC, Tbilisi, Georgia), in the course of attendance of patients to clinics.

Screening:

A comprehensive medical history will be ascertained by the study doctor. All patients will have a complete physical examination and laboratory evaluation. Patients with confirmed COVID-19 diagnosis based on positive SARS-Cov-2 test which will be assessed for eligibility.

Study information:

An information about the study in included in patient written consent and will be handed out to each subject. Before any study related procedures are initiated, all objectives, methods and potential hazards will be explained verbally to the subject by the investigator in Georgian language. The subject will be given sufficient opportunity to ask questions about study details and allowed time to consider the information provided. The subject information will clearly state that the subjects are completely free to enter or not to enter the study, or to withdraw from it whenever they want without negative consequences. Subjects will be informed that personal data will be treated with absolute confidentiality.

Informed consent:

All subjects have to give their written consent before taking part in the study. The Informed Consent Form must be dated and personally signed by each subject. The Principal Investigator (or designee) must store the original, signed Informed Consent Form. A copy of the Informed Consent Form must be given to the subject.

Schedule of examinations and procedures:

Day 1 (Visit 1. Screening, Baseline): Eligibility check /Information, Informed consent, Clinical examination, Allocation to intervention, Treatment, Lab Tests (COVID-19 PCR test, Blood serum cytokin IL-6 , D-Dimer, C-reactive protein, Cognitive performance test, Tests for anxiety-depression, assessment of Long COVID symptoms, Physical activity.

Day 7 (Visit 2): Clinical examination, Treatment, Lab Tests (Blood serum cytokin IL-6 , D-Dimer, C-reactive protein, Cognitive performance test, Tests for anxiety-depression, assessment of Long COVID symptoms, Physical activity, Adverse events.

Day 14 (Visit 3): Clinical examination, Treatment, Lab Tests (COVID-19 PCR test, Blood serum cytokin IL-6 , D-Dimer, C-reactive protein, Cognitive performance test, Tests for anxiety-depression, assessment of Long COVID symptoms, Physical activity, Adverse events, Drug intake accountability.

Day 21 (Visit 4, Follow up): Clinical examination, Lab Tests (Blood serum cytokin IL-6 , D-Dimer, C-reactive protein, Cognitive performance test, Tests for anxiety-depression, assessment of Long COVID symptoms, Physical activity, Adverse events.

Days 1, 3, 5, 7, 9, 11, 14, 21: Patient self-assessment of Long COVID symptoms, Physical activity and body temperature

During the visit 1, the investigator informs prospective participants regarding the test compound, the aims and nature of the study, and offers the opportunity of participation.

The investigator hands over the study diary - patient's self-assessment forms and Instruction to the participants and explains how to use it. The log contains questionaries, which should be filled in during the study.

Participants fill inn all questionnaires form under guidelines and with help of the Investigator. The investigator scores participants on the anxiety and depression using HAM-A, and HADS inventories. Patients provides blood samples for laboratory analysis and complete d2-test for attention and memory. After completion of all screen and baseline procedures, and after assuring that all study entry inclusion and exclusion criteria are met, patients sign the informed consent form. After that they will be randomly assigned to double-blind treatment with either ADAPT-232, 60 ml daily, or placebo and receive then package with investigational product.

Follow up Study Visits 2-4: Patients will then return for follow up study visits at weeks 2, 3 and 4. Each patient will be evaluated by the study doctor to assess the presence and severity of symptoms.

Patient will provide blood samples for laboratory testing and the study doctor will perform the d2-test HAM-A and HADS ratings. The study doctor will obtain a detailed safety profile of all adverse events including the dates of occurrence, severity of the event, and relationship to study medication (i.e., definite, probable, possible, unrelated). Patients will be specifically instructed by the study doctor not to use these agents during the trial. At each study visit, vital signs and weight will be obtained by the study coordinator (or a research nurse). Finally, the amount of oral solution (drug) record will be obtained by doctor.

After visit 3 (two weeks drug administration), no treatment is administered for one week.

On the last visit 4, patients will provide blood samples for laboratory testing and the study doctor will perform the d2-test HAM-A and HADS ratings and collects the study diary, and fill-in the Unused oral solution as well as the empty bottles are gathered. In case the subject does not report unwanted events, the investigator asks about side effects.

Criteria for discontinuation:

The study may be discontinued by participants at any time. Specific reasons for discontinuation are:

voluntary discontinuation by participants without any prejudice to further treatment, safety reasons as judged by the Investigator, severe non-compliance to the protocol as judged by the Investigator, incorrect enrolment i.e. participants do not meet the required inclusion/exclusion criteria.

Procedures for discontinuation:

Participants who discontinue after receiving the treatment will be deblinded and asked to deliver the remaining liquid to the investigator. All individuals will be asked about the reason(s) for their discontinuation and the presence of any adverse events.

Procedures for handling incorrectly enrolled participants:

Individuals not meeting inclusion/exclusion criteria for the study should, under no circumstances, be enrolled into the study - there can be no exception to this rule. Individuals that do not meet study criteria and are enrolled by mistake, incorrectly randomized, or subsequently fail to meet criteria for the study should return for the procedures and assessments to the study site.

Treatment compliance:

Participants are asked to take their daily dose of 60 ml oral solution. Participants will be questioned about their overall compliance with the study protocol upon their visits and the remaining tablets will be counted by the study personnel. Compliance will be monitored by the doctor. He will check patients' records in a special form which will be attached to Case Report Form (Appendix 8). Doctor will check overall compliance with the study protocol upon their visits and the remaining liquid will be measured by a measuring cylinder at the end of the study.

Data management plan (DMP):

All data will be handled in accordance with the study's Data Management Plan. The Data Management Plan (DMP) are developed by the CRO. Staff at the study that are involved in the data handling process are trained by their respective data manager according to the DMP.

Core data management activities will be carried out in a standardized manner and are documented properly. DMP describes the complete data handling process in the study.

It contains information about the following aspects: structure of the study database, data flow, handling of Case Report Forms, monitoring, data entry, data validation activities, database lock, activities assuring data security and backup, query management, correct documentation, further applicable documents, clarification of responsibilities. Emerging problems with and deviations from the DMP will to be reported to the CRO.

Monitoring:

The monitoring of this study will be performed in accordance with the principles of Good Clinical Practice (GCP) as laid out in the International Conference on Harmonisation (ICH) document "Good Clinical Practice: Consolidated Guideline". The monitoring includes, whether all study activities, including documentation and reporting are in accordance with the applicable SOPs, the study protocol and legal requirements. Monitoring takes place regularly and will be carried out by the Sponsor and includes source data verification. After completion of a monitoring visit, a report containing a description of the monitoring activities and their results is written.

Source data verification:

The Study Monitor is given direct access to source data for data verification. Source data are randomly checked for completeness and plausibility. Moreover, in case of paper-based source data that are also stored electronically data are also checked for entry errors. That is, the data-entries are compared with the paper version to check for transcription errors and omissions.

Audits and inspections Authorized representatives of Swedish Herbal Institute Research and Development AB, a regulatory authority or an ethical review board (ERB) may visit the study sites to perform audits or inspections, including source data verification. The purpose of such an audit or inspection is to systematically and independently examine all study-related activities and documents to determine whether they were performed in accordance to the protocol, GCP guidelines and any applicable regulatory requirements. These activities include the study procedure, data recording, management, analysis and reporting. After termination of the audit or inspection, main topics and findings are documented in a report. The Principal Investigator (or designee) should contact the Sponsor immediately if contacted by a regulatory agency about an inspection at his or her center.

Changes to the protocol:

Study procedures will not be changed without the mutual agreement of the Investigator and Sponsor. If it is necessary for the study protocol to be amended, the amendment and/or a new version of the study protocol must be notified and approved by the Sponsor before implementation. Local requirements must be followed.

Case report forms (CRF):

All information collected during the study will be documented independently for each subject in standardized paper Case Report Forms (CRFs) which are marked with a personal subject identification number. Data should be recorded legibly onto the CRFs in blue or black ballpoint pen. Correction fluid or covering labels must not be used. Standardized CRFs are created by the CRO and distributed to the Sponsor and each participating study site.

Data from the completed pCRFs will be entered onto National Family Medicine center clinical study database and validated under direction of the data manger. The data base should follow for reconciliation of serious adverse events (SAEs) by Swedish Herbal Institute Research and Development AB drug safety department. Any missing, impossible or inconsistent recordings in the pCRFs will be referred back to the Investigator using Data Query Forms and be documented for each individual before clean file status is declared.

Source data verification will be done by checking printouts of entered data against source data (i.e., laboratory results, questionnaires). Later questions and corrections will be noted and verified by the Investigator. Any missing, impossible or inconsistent entries in the database (or pCRF) will be referred back to the Investigator using data query forms, and be documented for each individual before clean file status is declared.

Data processing and analyses:

Intention-to-Treat analyses of data will take place after termination of the study and laboratory analyses. Data will be entered twice, and subsequently compared and cleaned for verification of correct input using the Excel and Prizm programs.

Handling of subjects' information:

Subjects' data are handled confidentially. The original data are only accessible for the Investigator. Subjects' data are encrypted after the study. Pseudonymized data can be transferred to the Sponsor. Original data is stored securely at NFMTC for ten years.

Statistical Methods and Determination of Sample Size

Statistical and analytical plans The clinical data at each visit will be recorded using a standardized clinician assessment form (case reports form - CRF) and collected in an Excel database, which will be used for further analysis using statistical software GraphPad (San Diego, CA, USA) Prism software (version 3.03 for Windows).

The approach for analysis of the primary and secondary outcomes from this study will be similar. To assess whether the treatment groups are similar at baseline, the mean outcomes will be compared at baseline for subjects who receive ADAPT-232 vs. placebo by the Student's parametric independent-measures t-test (variables with normal distribution) or Mann-Whitney non-parametric test, depending on results of normality test.

Analysis of changes within treatment groups during the study (Visits 1,2,3 and 4) will be performed by:

* One-way, repeated measures ANOVA (variables with normal distribution),
* Friedman test for repeated several measures (nonparametric data),

Assessment of efficacy of study medications will be achieved by comparison of mean changes from the baseline (differences before and after treatment of every single patient) between groups using two-way between-within ANOVA in which an interaction effect indicates a different response over time between the two groups and would therefore signal a treatment effect, as well as by multiple comparison t-test (one unpaired test per row),

The primary end point was defined as the Duration of the Symptoms. Kaplan-Meier curves will be generated for all end points, and medians were calculated from those curves. The treatment arms will be compared by Mantel-Cox log-rank and Gehan-Breslow-Wilcoxon tests. The estimates of treatment hazard ratios based on log-rank tests and 95% CIs were calculated.

Intergroup comparison of number patients with particular symptoms will be assessed using the odds ratio (OR) statistics of endpoints according to Altman; A/B test of significance of differences of endpoints at 95% confidence, and z-statistic at 95% confidence of statistical significance.

The incidence of adverse events will compared across treatment groups for descriptive purposes and to identify possible differences in the safety profiles using the odds ratio (OR) statistics of endpoints according to Altman; A/B test of significance of differences of endpoints at 95% confidence; and z-statistic methods for categorical data https://www.medcalc.org/calc/odds_ratio.php

A statistical significance level of 5% was used in the Protocol approved by the health authorities. Statistical analysis will be performed on an intent-to-treat basis.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 patients with confirmed diagnosis based on positive SARS-Cov-2 test and the symptom of at least three of Long COVID-19 symptoms including: fatigue, headache, respiration problems (dyspnea or polypnea), sweat, cognitive disorders (attention, memory, anxiety and depression), loss of smell (anosmia) and taste (ageusia), cough, pain in joints. muscles and chest.
* Post COVID-19 patients discharged from Covid Hotels isolation, after hospitals and Intensive Care Unit (ICU) admission.
* Subjects must be under observation or admitted to a controlled facility or hospital (home quarantine is not sufficient).
* Able to take medication alone.
* Able to give informed consent.

Exclusion Criteria:

* Post COVID-19 patients discharged from Covid Hotels isolation, after hospitals and Intensive Care Unit (ICU) admission and Long Covid Symptoms longer that 3 months.
* Patient admitted already under invasive mechanical ventilation;
* Patient admitted with severe acute respiratory syndrome and diagnosed with an etiologic agent other than SARS-CoV-2;
* Renal failure requiring dialysis or creatinine ≥ 2.0mg/dl;
* Tube feeding or parenteral nutrition.
* Respiratory decompensation requiring mechanical ventilation.
* Uncontrolled diabetes type 2.
* Autoimmune disease.
* Pregnant or lactating women.
* Taking antibiotics for a reason other than COVID-19 at enrollment;
* Has a chronically weakened immune system (AIDS, lymphoma, chemo-radio- corticosteroid therapy, immunosuppressive pathology);
* Was treated with chemo-radio-corticosteroid therapy in the last 6 months;
* Has active cancer;
* Taking immunosuppressive drugs (e.g. anti-rejection treatment after organ transplant);
* Already participating in another clinical trial;
* Has any other condition that would prevent safe participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2021-11-11 (Actual); Study Completion 2021-12-26 (Actual)

PRIMARY OUTCOMES:
Duration of symptoms of Long COVID: | Change from baseline during the period of the treatment and follow up (from Day 1 to Day 14 and day 21 after randomization)
  Time (days) from randomization to symptoms disappear
Number of participants clinically recovered | Change from baseline during the period of the treatment and follow up (from Day 1 to Day 14 and day 21 after randomization)
  Number of participants without symptoms of Long COVID
Length of home stay/ sick listed | Change from baseline during the period of the treatment and follow up (from Day 1 to Day 14 and day 21 after randomization)
  Time (days) at home / sick listed
Severity of the Long COVID symptoms | Change from baseline during the period of the treatment and follow up (trough 21 days after randomization)
  Time from randomization to relief of total and individual Long COVID symptoms scores Patient will be assessed for changes in clinical signs: headache, fatigue, physical activity, depression and anxiety, anosmia, ageusia, hair loss, cough, fever, sweat, pain in muscles, chest, and joints. The medians and hazard ratio's will be measured and compared between groups)

SECONDARY OUTCOMES:
Hypercoagulation marker | Change from baseline during the period of the treatment and follow up (from Day 1 to Day 14 and day 21 after randomization)
  D-Dimer
Immune response marker | Change from baseline during the period of the treatment and follow up (from Day 1 to Day 14 and day 21 after randomization)
  IL-6 concentration in the serum (pg/ml).
Inflammatory marker | Change from baseline during the period of the treatment and follow up (from Day 1 to Day 14 and day 21 after randomization)
  C-reactive protein
Physical activity | Change from baseline during the period of the treatment and follow up (from Day 1 to Day 14 and day 21 after randomization)
  Assessed by Habitual Physical Activity Questionnaire Score
Cognitive performance score | Change from baseline during the period of the treatment and follow up (from Day 1 to Day 14 and day 21 after randomization)
  d2 - test of attention and memory.
Severity of anxiety and depression | Change from baseline during the period of the treatment and follow up (from Day 1 to Day 14 and day 21 after randomization)
  Severity of anxiety and depression assessed by Hospital Anxiety and Depression Scale (HADS)
Severity of anxiety | Change from baseline during the period of the treatment and follow up (from Day 1 to Day 14 and day 21 after randomization)
  Severity of anxiety assessed by Hamilton Anxiety Rating Scale

OTHER OUTCOMES:
Time to negative COVID-19 test | 14 days after randomization
  SARS-Cov-2 PCR test

CONTACTS AND LOCATIONS:
Overall Officials: Irina Karosanidze, PhD, MD, Principal Investigator — Director of National Family Medicine Training Centre
Locations (1):
- National Family Medicine Training Centre,, Tbilisi, Georgia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Panossian A, Brendler T. The Role of Adaptogens in Prophylaxis and Treatment of Viral Respiratory Infections. Pharmaceuticals (Basel). 2020 Sep 8;13(9):236. doi: 10.3390/ph13090236. PMID 32911682
- [Background] Brendler T, Al-Harrasi A, Bauer R, Gafner S, Hardy ML, Heinrich M, Hosseinzadeh H, Izzo AA, Michaelis M, Nassiri-Asl M, Panossian A, Wasser SP, Williamson EM. Botanical drugs and supplements affecting the immune response in the time of COVID-19: Implications for research and clinical practice. Phytother Res. 2021 Jun;35(6):3013-3031. doi: 10.1002/ptr.7008. Epub 2020 Dec 29. PMID 33373071
- [Background] Narimanian M, Badalyan M, Panosyan V, Gabrielyan E, Panossian A, Wikman G, Wagner H. Impact of Chisan (ADAPT-232) on the quality-of-life and its efficacy as an adjuvant in the treatment of acute non-specific pneumonia. Phytomedicine. 2005 Nov;12(10):723-9. doi: 10.1016/j.phymed.2004.11.004. PMID 16323290
- [Background] Lopez-Leon S, Wegman-Ostrosky T, Perelman C, Sepulveda R, Rebolledo PA, Cuapio A, Villapol S. More than 50 Long-term effects of COVID-19: a systematic review and meta-analysis. medRxiv [Preprint]. 2021 Jan 30:2021.01.27.21250617. doi: 10.1101/2021.01.27.21250617. PMID 33532785
- [Background] Tenforde MW, Kim SS, Lindsell CJ, Billig Rose E, Shapiro NI, Files DC, Gibbs KW, Erickson HL, Steingrub JS, Smithline HA, Gong MN, Aboodi MS, Exline MC, Henning DJ, Wilson JG, Khan A, Qadir N, Brown SM, Peltan ID, Rice TW, Hager DN, Ginde AA, Stubblefield WB, Patel MM, Self WH, Feldstein LR; IVY Network Investigators; CDC COVID-19 Response Team; IVY Network Investigators. Symptom Duration and Risk Factors for Delayed Return to Usual Health Among Outpatients with COVID-19 in a Multistate Health Care Systems Network - United States, March-June 2020. MMWR Morb Mortal Wkly Rep. 2020 Jul 31;69(30):993-998. doi: 10.15585/mmwr.mm6930e1. PMID 32730238
- [Background] Rogers JP, Chesney E, Oliver D, Pollak TA, McGuire P, Fusar-Poli P, Zandi MS, Lewis G, David AS. Psychiatric and neuropsychiatric presentations associated with severe coronavirus infections: a systematic review and meta-analysis with comparison to the COVID-19 pandemic. Lancet Psychiatry. 2020 Jul;7(7):611-627. doi: 10.1016/S2215-0366(20)30203-0. Epub 2020 May 18. PMID 32437679
- [Background] Panossian AG, Efferth T, Shikov AN, Pozharitskaya ON, Kuchta K, Mukherjee PK, Banerjee S, Heinrich M, Wu W, Guo DA, Wagner H. Evolution of the adaptogenic concept from traditional use to medical systems: Pharmacology of stress- and aging-related diseases. Med Res Rev. 2021 Jan;41(1):630-703. doi: 10.1002/med.21743. Epub 2020 Oct 25. PMID 33103257